CLINICAL TRIAL: NCT04821245
Title: Defining Normal Postoperative Magnetic Resonance Imaging and Muscle Enzyme Levels After Total Knee Arthroplasty Associated With Continuous Adductor Canal Block
Brief Title: Defining Normal Postoperative Magnetic Resonance Imaging After Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Benaroya Research Institute (Other)
Collaborators: Washington State Society of Anesthesiologists (Other)
Responsible Party: Principal Investigator, Joseph M. Neal, Affiliate Investigator, Benaroya Research Institute
Other Study IDs: BRI IRB18-008
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Results first posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Local Anesthetic Complication; Local Anesthetic Drug Adverse Reaction
Keywords: Myotoxicity; Myositis; Magnetic resonance imaging; Creatine phosphokinase; Aldolase
MeSH Terms: conditions — Myotoxicity; Myositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
The aim of this study was to describe the postoperative "baseline" magnetic resonance imaging (MRI) appearance of the ipsilateral thigh musculature after total knee arthroplasty (TKA). The secondary aim was to describe baseline muscle enzyme levels under the same clinical scenario. Neither of these measures have been reported previously.

DETAILED DESCRIPTION:
* In 2016, 3 sentinel cases of presumed local anesthetic-induced myotoxicity were reported after TKA with associated continuous adductor canal block (CACB) analgesia. The diagnosis was made based on its consistency with animal and human descriptions of local anesthetic myotoxicity, including: a) exposure to local anesthetic, b) delayed symptom onset after a period of normal recovery, c) rapid development of profound muscle flaccidity, and d) complete to partial recovery of motor function after weeks to months. MRIs obtained in these patients showed diffuse intra- and inter-muscular edema (inflammation) of the ipsilateral thigh, which was believed to support the presumptive diagnosis. However, because baseline MRI appearance of upper leg muscles has never been described for this clinical scenario, it is possible that the MRI scans represented "normal, baseline" appearance.
* This case series intended to prospectively describe postoperative MRI appearance in a cohort of asymptomatic volunteer patients that underwent uncomplicated TKA/CACB. In addition, because obtaining biomarkers of muscle injury might also be a reasonable diagnostic step, we sought to measure preoperative and postoperative creatine phosphokinase (CPK) and aldolase levels.
* MRI scans were read by 5 board-certified musculoskeletal radiologists masked to the study's purpose. Grading was done using a standard grid that facilitated systematic evaluation of various regions within the upper leg. At least 3 of 5 radiologists were required to declare edema as present within a given region of the leg.
* Only those volunteer patients that presented a normal postoperative course, i.e., had no unexpected leg muscle weakness, were entered into the study. As such, the MRI and muscle enzyme analysis results had no impact on the volunteer patients' clinical outcome or management. This was a prospective, observational/descriptive case series. There was no control group and we did not intend to investigate issues of cause-and-effect.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for unilateral primary TKA with CACB
* TKA and early recovery was uncomplicated (no evidence of unexpected leg weakness)

Exclusion Criteria:

* Contraindication to spinal anesthesia or adductor canal-based analgesia
* History of muscle wasting or related disease
* History of autoimmune disorders that may affect muscles
* History of neurologic condition affecting the lower extremities
* Contraindications to MRI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Volunteer patients of various age and sex
  * Number of volunteers and diagnostic studies determined by available grant monies
  * Volunteers were drawn from a population presenting for unilateral primary TKA performed by 1 of 2 orthopedic surgeons in a single institution
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Neal, MD, Principal Investigator — Benaroya Research Center at Virginia Mason Medical Center
Locations (1):
- Benaroya Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified raw data in Excel format may be obtained from Joseph M. Neal, MD upon request.
Time Frame: March 2021 through March 2026
Access Criteria: Upon request

REFERENCES:
- [Background] Neal JM, Salinas FV, Choi DS. Local Anesthetic-Induced Myotoxicity After Continuous Adductor Canal Block. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):723-727. doi: 10.1097/AAP.0000000000000466. PMID 27662067
- [Background] Neal JM, Salinas FV, Choi DS. Reply to Dr Kelly et al. Reg Anesth Pain Med. 2017 May/Jun;42(3):414. doi: 10.1097/AAP.0000000000000574. No abstract available. PMID 28419048
- [Background] Hussain N, McCartney CJL, Neal JM, Chippor J, Banfield L, Abdallah FW. Local anaesthetic-induced myotoxicity in regional anaesthesia: a systematic review and empirical analysis. Br J Anaesth. 2018 Oct;121(4):822-841. doi: 10.1016/j.bja.2018.05.076. Epub 2018 Aug 8. PMID 30236244
- [Derived] Mahyar L, Neal JM, Blackmore CC, Jackson DW, Hanson NA, MacDonald KM, Warren D, Verdin PJ. MRI and muscle enzymes do not support the diagnosis of local anesthetic myotoxicity: a descriptive case series. Reg Anesth Pain Med. 2021 Aug;46(8):679-682. doi: 10.1136/rapm-2021-102772. Epub 2021 May 31. PMID 34059556

RESULTS

PARTICIPANT FLOW:
Recruitment Details: * Tertiary care medical center
  * December 2018 through August 2019
  * Potential volunteers were contacted by the principal investigator at least 24 hours prior to their surgery. Informed consent was obtained at this point.
  * Volunteers could decline to proceed at any point from initial informed consent through MRI scan or final blood draw
Pre-assignment Details: -Volunteer patients only entered the study if they showed no signs of unexpected ipsilateral upper leg weakness prior to drawing blood samples or obtaining MRI scans
Groups:
- Single Cohort: All volunteer patients
Period: Overall Study
Arm/Group | Single Cohort
Started | 36
Completed | 27
Not Completed | 9
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1
Not completed — Protocol Violation | 5

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: All enrolled subjects
Arm/Group | Overall Study
Number analyzed (Participants) | 27
Age, Continuous [Mean (Full Range); unit: years] | 62 [46 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Mean (Full Range); unit: kg] | 89 [59 to 134]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Edema
Description: Regions of the ipsilateral thigh were defined by muscle group, neuromuscular bundle, subcutaneous tissue, or inter-muscular fascial layers. Five board-certified musculoskeletal radiologists analyzed the scans for presence of edema. Edema was considered present if judged to be so by at least 3 of the 5 radiologists.
Time Frame: 1-2 days postoperative
Population: Participants that underwent postoperative MRI scan of operated leg
Measure: Number; unit: participants
Groups:
- Participants Undergoing MRI: Number of Participants with Edema
Arm/Group | Participants Undergoing MRI
Number analyzed (Participants) | 12
participants | 12

2. Secondary Outcome: Postoperative Muscle Enzyme Levels
Description: Participants with Postoperative Creatine Phosphokinase (CPK) or Aldolase levels above the upper limit of normal
Time Frame: Sample was drawn the morning after surgery
Population: Participants with CPK levels 12% to 111%, and aldolase levels, in excess of high normal values
Measure: Count of Participants; unit: Participants
Groups:
- CPK Analysis: CPK Levels Above High Normal
- Aldolase Analysis: Aldolase Levels Above High Normal
Arm/Group | CPK Analysis | Aldolase Analysis
Number analyzed (Participants) | 19 | 19
Participants | 5 | 0

ADVERSE EVENTS:
Time Frame: 10 days. Participant was evaluated at the time of the incident and twice during the 10 days thereafter.
Groups:
- MRI Appearance: Volunteers undergoing MRI examination
Arm/Group | MRI Appearance
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 1/13
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MRI Appearance (N=13)
Warmth around adductor canal catheter during MRI (Musculoskeletal and connective tissue disorders) | 1 (1) — As described above - mild, vague warmth around catheter at start of MRI, which was subsequently cancelled. The warmth resolved quickly and the patient was not harmed.

LIMITATIONS AND CAVEATS:
This case series aimed to describe MRI appearance and muscle enzyme levels presented under the same clinical conditions as the 3 sentinel cases of presumed local anesthetic myotoxicity after TKA/CACB. This descriptive design was not intended to sort cause-and-effect (that is, the relative role of surgery, pneumatic tourniquet, local anesthetic, etc.) in causing muscular edema or raising enzyme levels.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: w/o statistical comment (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/45/NCT04821245/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (specific comment) (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/45/NCT04821245/SAP_001.pdf
  • Informed Consent Form (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/45/NCT04821245/ICF_002.pdf